CLINICAL TRIAL: NCT06851845
Title: Clinical Outcomes of C3 Glomerulopathy and IC-MPGN in Russia: Hybrid Retrospective - Prospective Study
Acronym: CRYSTAL
Status: Not yet recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023B1RU01
Record Dates: First submitted 2025-02-12; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Kidney Diseases
Keywords: glomerulopathy
MeSH Terms: conditions — Kidney Diseases | interventions — Adrenal Cortex Hormones; Cyclophosphamide; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- C3 glomerulopathy: Diagnosis of primary C3G confirmed by the results of morphological and clinical studies.
  Interventions: Other: No intervention
- Immune-complex membranoproliferative glomerulonephritis: Diagnosis of primary IC-MPGN confirmed by the results of morphological and clinical studies.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will receive medical care in accordance with the routine practice of disease treatment
  Other Names: Treatment includes the following options:; ACEi/ARB alone; ACEi/ARB + corticosteroids; ACEi/ARB + MMF; ACEi/ARB + SGLT2i; ACEi/ARB + MMF + corticosteroids; ACEi/ARB + cyclophosphamide; Corticosteroids alone; MMF alone; Cyclophosphamide alone; Corticosteroids + MMF; Rituximab; Anticomplement therapy; Other immunosuppressants

SUMMARY:
The study is planned to study specificity of the clinical course and treatment outcomes of C3 glomerulopathy (C3G) and Immune-complex membranoproliferative glomerulonephritis (IC-MPGN) in patients aged under 18 years and 18 years and older in the Russian population in 2025-2028. The primary objective of the study is to estimate the frequency of complete or partial remission 12 months after morphological verification of the diagnosis. Assessment of demographic, clinical and laboratory, morphological characteristics at diagnosis and their relationship with the disease outcomes, primarily the disease progression and development of chronic renal failure, will allow assessing the efficacy of treatment used in real clinical practice, disease prognosis and factors associated with unfavourable outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign informed consent form. If the patient is under 18 years of age, the parent or legally acceptable representative of the child/adolescent who can participate in this study also signs the consent form.
2. Diagnosis of primary C3G or IC-MPGN confirmed by the results of morphological and clinical studies.
3. The results of serum creatinine level, proteinuria determination obtained not earlier than 4 weeks before the kidney biopsy
4. Index date (kidney biopsy) not earlier than March 2024 and not later than 11 months before signing the ICF
5. The estimated baseline GFR (using the CKD-EPI formula for persons aged over 18 years and the modified Schwarz formula for children) or the measured GFR is ≥30 mL/min per 1.73 m2.

Exclusion Criteria:

1. Patients participating in a clinical trial with the investigational product.
2. Patients with monoclonal gammopathies (myeloma, B-cell lymphoma/lymphocytic leukemia, lymphoplasmacytoma)
3. Patients with systemic autoimmune diseases and vasculitis (systemic lupus erythematosus, systemic sclerosis, dermatomyositis, mixed connective tissue disease, Sjogren syndrome, Henoch-Schönlein purpura, ANCA vasculitis, cryoglobulinemia)
4. Patients with current or recent infections (viral hepatitis B, viral hepatitis C, infective endocarditis or sepsis, infected ventriculoatrial shunts, abscesses, meningococcal and other bacterial infections, protozoan infections)
5. Patients with any clinically significant acute disease within 30 days prior to kidney biopsy
6. Clinically significant concomitant kidney disease
7. Treatment with pegcetacoplan

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will recruit adults (aged 18 years and older) and pediatric patients (legally acceptable representatives) with biopsy-confirmed diagnosis of primary C3G or idiopathic IC-MPGN in the period from March 2024 to February 2027, who will meet the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of patients with overall (complete + partial) remission following the standard therapy in Russia | 12 months
  Complete response is defined as proteinuria <0.5 g/24 h with stable eGFR (less than 20% decline in eGFR from baseline without the need for renal replacement therapy).
  Partial response is defined as reduction of proteinuria at stable eGFR (no decrease of >20% of baseline value): >50% (from baseline) (in those with proteinuria <3.5 g/day or >3.5 g/day but without nephrotic syndrome (NS)) OR in ≥50% from baseline accompanied by a regression of NS (NS <3.5 g/day and blood albumin ≥30 g/L).

SECONDARY OUTCOMES:
Number and proportion of patients with complete remission | 6 months; 12 months
  Complete remission was defined as proteinuria <0.5 g/24 h with a stable eGFR (less than 20% decline in eGFR from baseline without the needs for renal replacement therapy).
Number and proportion of patients with partial remission | 6 months; 12 months
  Partial remission was defined as a reduction in proteinuria at stable eGFR (no decrease of >20% of baseline): >50% (from baseline) (in those with proteinuria <3.5 g/day or >3.5 g/day but without nephrotic syndrome (NS)) OR in ≥50% from baseline accompanied by a regression of NS (NS: <3.5 g/day and blood albumin ≥30 g/L)
Number and proportion of patients with relapse | 6 months; 12 months
  Clinical relapse was defined as a proteinuria >3.5 g/24h after achieving complete remission or, in those with partial remission, as an increase of proteinuria >50% compared with the lowest value during remission with recurrence of NS
Number and proportion of patients with progression | 6 months; 12 months
  Composite progression defined as 40% eGFR decline from the baseline and/or eGFR <15 mL/min per 1.73 m2 and/or renal replacement therapy
Number and proportion of patients with progression to end-stage kidney disease | 6 months; 12 months
  Number and proportion of patients with progression to end-stage kidney disease from index-date up to 12 months
Number and proportion of died patients | 6 months; 12 months
  Number and proportion of patients who died from index date up to 12 months
Time to start of maintenance dialysis | 6 months; 12 months
  Time in months from index date to start of maintenance dialysis
Time from the diagnosis date to the start date of dialysis | 6 months; 12 months
  Time in months from the diagnosis date to the start date of dialysis
Time from the start date of treatment to the start date of dialysis | 6 months; 12 months
  Time in months from first treatment date to the start date of dialysis
Time from the diagnosis date to transplantation | 6 months; 12 months
  Time in months from the diagnosis date to transplantation
Time from the diagnosis date to the date of complete remission | 6 months; 12 months
  Time in months from the diagnosis date to the date of complete remission
Time from the diagnosis date to the date of partial remission | 6 months; 12 months
  Time in months from the diagnosis date to the date of partial remission
Time from the diagnosis date to the date of overall remission (complete and partial remission) | 6 months; 12 months
  Time in months from the diagnosis date to the date of overall remission (complete and partial remission)
Time to progression | 6 months; 12 months
  Time in months from the diagnosis date to progression
Number and proportion of patients with a) an increase in eGFR by ≥15% from the baseline; b) decrease in eGFR by ≥15% from the baseline; c) stable eGFR (change up to 15%) | 6 months; 12 months
  Number and proportion of patients with a) an increase in eGFR by ≥15% from the baseline; b) decrease in eGFR by ≥15% from the baseline; c) stable eGFR (change up to 15%) from index date up to 12 months
Time to 30%, 40% and 50% decline in eGFR | 6 months; 12 months
  Time in months from index date to 30%, 40% and 50% decline in eGFR
Number and proportion of patients with proteinuria >1 g/24 h and eGFR ≥30 mL/min per 1.73 m2 | 6 months; 12 months
  Number and proportion of patients with proteinuria >1 g/24 h and eGFR ≥30 mL/min per 1.73 m2 from index date up to 12 months
Number and proportion of patients with nephrotic syndrome | 6 months; 12 months
  Number and proportion of patients with nephrotic syndrome from index date up to 12 months
Demographic and clinical characteristics of patients with primary C3G (cohort 1), IC-MPGN (cohort 2), and overall | Baseline
  Number and proportion of patients by age, gender, BMI, BSA, family history of kidney disease, transplant status, blood pressure, laboratory markers: serum creatinine level (µmol/L), eGFR, urinary blood cell (RBCs/hpf), proteinuria (g/24h), serum albumin (g/L); eGFR rate of change; chronic kidney disease (CKD) stage; proteinuria ≥1 g/24 h AND eGFR ≥30 mL/min per 1.73 m2
Number of patients by morphologically verified disease form in patients with primary C3G (cohort 1), IC-MPGN (cohort 2), and overall | Baseline
  Morphologically verified disease form: DDD (subject to electron microscopy), C3GN (subject to electron microscopy), C3G (in the absence of informative electron microscopy data), IC-MPGN.
Number of patients with presence of serum complement markers, serum factor H, rare genetic variants | Baseline
  Number of patients with presence of serum complement markers (C3, C4, CH50, C5a), serum factor H, rare genetic variants at baseline
Number and proportion of patients stratified by treatment sequence and specific regimen of treatment | Baseline; 6 months; 12 months
  Number and proportion of patients stratified by treatment sequence and specific regimen of treatment
Number and proportion of patients that discontinued a specific regimen of treatment at each line of therapy at any time during follow-up and reason for discontinuation for each cohort | Baseline; 6 months; 12 months
  Number and proportion of patients that discontinued a specific regimen of treatment at each line of therapy at any time during follow-up and reason for discontinuation for each cohort
Number of exposed doses for non-continuous treatments (e.g., pulse therapy, rituximab infusion) in each cohort | Baseline; 6 months; 12 months
  Number of exposed doses for non-continuous treatments (e.g., pulse therapy, rituximab infusion) in each cohort
Number of patients by qualitative, semi-quantitative and quantitative scores of active and chronic lesions | Baseline
  1. mesangial proliferation (% of glomeruli),
  2. endocapillary hypercellularity (% of glomeruli),
  3. membranoproliferative morphology (thickening and/or double contouring of the capillary basement membranes),
  4. leukocyte infiltration,
  5. proportion of completely intact glomeruli (%)
  6. proportion of cellular (%), fibrous (%), fibrocellular (%) crescents,
  7. fibrinoid necrosis,
  8. interstitial infiltration,
  9. interstitial fibrosis (%),
  10. tubular atrophy (%),
  11. global and segmental glomerulosclerosis (quantitatively, % of all glomeruli)
  12. arteriosclerosis and arteriolosclerosis
Number of patients with signs of thrombotic microangiopathy in the biopsy specimen | Baseline
  Number of patients with signs of thrombotic microangiopathy in the biopsy specimen at baseline
Number of patients with acute tubular necrosis | Baseline
  Number of patients with acute tubular necrosis at baseline
Number of patients with presence of C1q, IgA, IgM, IgG, C3, kappa chain, lambda chain deposits | Baseline
  Number of patients with presence of C1q, IgA, IgM, IgG, C3, kappa chain, lambda chain deposits at baseline
Patient-reported outcomes for C3G (cohort 1), IC-MPGN (cohort 2), and overall | 12 months
  1. Descriptive adherence data based on question score
  2. Patient-reported outcomes, SF-36 (RAND)
Number of patients (%) with adverse events/serious adverse events by treatment option | 12 months
  Number of patients (%) with adverse events/serious adverse events by treatment option from index date up to 12 months
Change from baseline of systolic and diastolic blood pressure (BP) in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline of systolic and diastolic blood pressure (BP) (with percentiles for children) at 6 and 12 month
Change from baseline serum creatinine level (µmol/L) in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline serum creatinine level (µmol/L) at 6 and 12 months
Change from baseline estimated glomerular filtration rate (eGFR) in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline estimated glomerular filtration rate (eGFR) at 6 and 12 months
Change from baseline eGFR rate of change over time (eGFR slope) in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline eGFR rate of change over time (eGFR slope) at 6 and 12 months
Change from baseline chronic kidney disease (CKD) stage (number of patients, %) in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline chronic kidney disease (CKD) stage (number of patients, %) at 6 and 12 months
Change from baseline red blood cell count in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline red blood cell (RBC) count at 6 and 12 months
Change from baseline RBC casts in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline RBC casts at 6 and 12 months
Change from baseline daily proteinuria (proteinuria in g/24 hours) in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline daily proteinuria (proteinuria in g/24 hours) at 6 and 12 months
Change from baseline proteinuria >1 g/24 h in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline proteinuria >1 g/24 h at 6 and 12 months
Change from baseline eGFR ≥30 mL/min per 1.73 m2 in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline eGFR ≥30 mL/min per 1.73 m2 at 6 and 12 months
Change from baseline number of patients with nephrotic syndrome (%) in patients with C3G (cohort 1), IC-MPGN (cohort 2), and overall | 6 months; 12 months
  Change from baseline number of patients with nephrotic syndrome (%) at 6 and 12 months

IPD SHARING:
Plan to Share IPD: No